CLINICAL TRIAL: NCT02570932
Title: Intrathecal Administration (Pattern 100/3) of Expanded Autologous Adult Bone Marrow Mesenchymal Stem Cells in Established Chronic Spinal Cord Injuries
Brief Title: Administration of Expanded Autologous Adult Bone Marrow Mesenchymal Cells in Established Chronic Spinal Cord Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Jesús Vaquero Crespo, M.D., Principal Investigator, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CME-LEM3; 2014-005613-24 (EudraCT Number)
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Spinal Cord Injury
Keywords: Adult Autologous Bone Marrow Mesenchymal Cells Expanded; chronic spinal cord injury (SCI)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Mesenchymal Bone Marrow Cell (Experimental): All patients will be treated with the same treatment: Adult Autologous Mesenchymal Bone Marrow expanded Stem Cell (CME)
  Pharmaceutical form: Suspension in autologous plasma cell Route of administration: Intrathecal in subarachnoid space by lumbar puncture. Dose: Total dose of 300 x 106 CME, given in 3 injections of 100 x 106 CME, at intervals of 3 months between each administration.
  Interventions: Biological: Autologous Mesenchymal Bone Marrow Cell

INTERVENTIONS:
Biological: Autologous Mesenchymal Bone Marrow Cell — Suspension in autologous plasma cell of Adult mesenchymal stem cells expanded autologous bone marrow.
  Route of administration: Intrathecal in subarachnoid space by lumbar puncture.Total dose of 300 x 106 CME, divided in 3 injections of 100 x 106 CME, with intervals of three months between each administration

SUMMARY:
The purpose of this study is to analyze the potential clinical efficacy of intrathecal administration, in the subarachnoid space, of in vitro expanded autologous adult bone marrow mesenchymal stem cells in the treatment of patients with established chronic spinal cord injury (LEM).

DETAILED DESCRIPTION:
This is a clinical trial phase II, single-center, non-randomized, uncontrolled, open prospective follow-up of a cohort of patients with chronic spinal cord injury.

Patients are treated with repeated administrations of in vitro expanded autologous adult bone marrow mesenchymal stem cells.

The expanded cells are administered in the subarachnoid space by lumbar puncture. The minimum duration of the follow-up period for each patient is 10 months after the first administration.

The study duration is 24 months, that include recruiting, treatment and follow period for all patients. For each patient at the first day will be administered the first cellular doses, then 3 doses will be administrated every 3 months. At the end of the clinical trial, a completed check of all obtained parameters will be performed.

It is considered Day 1 for each patient the first day of the first cell administration. The remaining 2 doses will be administered at intervals of 3 months from the first administration (of the treatment period after, months 4 and 7). At the end of the study will be performed a full assessment of the variables collected along the study trial.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord injury (Level A, B, C or D in ASIA scales), clinically stable for at least 6 months prior to study start.
2. Previous studies of Neurophysiology, MRI and Urology to allow useful baseline, in order that they can be compared with the same scans following treatment, and to obtain objective data of potential efficacy.
3. Age between 18 and 70 years.
4. Men and women of childbearing age must compromise to use contraceptives from the time at which the removal of cells from the bone marrow is performed until 6 months after the Mesenchymal Stem Cells (MSC) last administration by lumbar puncture.
5. Possibility of follow up and ability to perform ambulatory physical therapy throughout all treatment period.
6. Written informed consent, according to the law in force.
7. Hematologic, creatinine, Serum glutamic oxaloacetic transaminase (SGOT) and Serum glutamic pyruvic transaminase (SGPT) parameters, within the normal range, according to laboratory standards. However, slight modifications that are considered significant in the context of treatment to be performed, according to the criterion of the research team, are accepted.

Exclusion Criteria:

1. Age below 18 years or above 70.
2. Pregnancy or lactation.
3. Current neoplastic disease or in the previous 5 years (diagnosed or treated).
4. Patients with systemic disease that represents an added risk to treatment.
5. Alterations in the genetic study performed to discard risk cell transformation in the expansion process.
6. Patients with doubts about possible cooperation in the maintenance physical therapy or in the controls carried out during the study
7. Neurodegenerative disease added.
8. History of substance abuse, psychiatric disease or allergy to protein products used in the process of cell expansion.
9. Positive serology for HIV and syphilis.
10. Active Hepatitis B or Hepatitis C, according to serology analysis.
11. If in the opinion of the researcher there is some other reason why the patient is not considered candidate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Changes in IANR-SCIFRS score are considerate for the motor and sensory functions evaluation. | from baseline until the end of the follow up period (24 months)
  Efficacy evaluation by measuring the change in motor and sensory functions by using the international Association of Neurorestoratology-Spinal Cord Injury Functional Rating Scale (IANR-SCIFRS). This scale includes 9 categories with 16 items in total (plus one optional category).
  The maximum possible score is 48; the lowest possible score is 0.

SECONDARY OUTCOMES:
Neurotrophic factors levels in Cerebrospinal fluid (CSF) and/ or Number of Adverse Events related to treatment | from baseline to 24 months
  The clinical evaluation of possible adverse effects is performed throughout the entire study duration and will be measured by descriptive analysis
Changes in PENN score are considerate for the motor and sensory functions evaluation | from baseline until the end of the follow up period (24 months)
  Efficacy evaluation by measuring the change in motor and sensory functions by using the Penn Spasm Frequency Scale that is Composed of 2-parts: the first is a self-report measure with items on 5-point scales developed to augment clinical ratings of spasticity and provides a more comprehensive assessment of spasticity
Changes in VAS score are considerate for quantification of pain | from baseline until the end of the follow up period (24 months)
  Efficacy evaluation by measuring the change in pain by using the visual analogue scale (VAS). The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks, depending on his feel of pain.
Changes in BDS score are considerate for the Assessment of the functional status | from baseline until the end of the follow up period (24 months)
  Efficacy evaluation by measuring the change in the Blepharospasm Disability Scale (BDS)
Changes in GEFFNER score are considerate for the Assessment of the functional status | from baseline until the end of the follow up period (24 months)
  Efficacy evaluation by measuring the change in the GEFFNER score

CONTACTS AND LOCATIONS:
Overall Officials: Jesús JV Vaquero Crespo, MD., Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda
Locations (1):
- Hospital Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data of participants will be shared with Authorities at the end of the Clinical development plan by the CTD (Common Technical Document). Results will be published in a scientific publication
Time Frame: Starting at CTD submission to authorities.
Access Criteria: Spanish competent authority.